CLINICAL TRIAL: NCT06249399
Title: The Effect Of Aerobic Exercise On Bladder Function And Lower Urinary Tract Symptoms In Women Who Has Diabetes Mellitus With Lower Urinary Tract Symptoms
Brief Title: The Effect of Aerobic Exercise on Lower Urinary System Symptoms in Women With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Collaborators: University of Gaziantep (Other); Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Bengisu Tüfekçi, Principal Investigator, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GİBTU-FP-BT-01
Record Dates: First submitted 2024-01-12; First posted 2024-02-08 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Lower Urinary Tract Symptoms; Diabetes Mellitus, Type 2
Keywords: Lower urinary tract symptoms; Diabetes Mellitus, Type 2; bladder; aerobic exercise; quality of life
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two groups: aerobic exercise group and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Group (Experimental): A behavioral treatment program will be applied to the patients. In addition, patients will be given submaximal aerobic exercise.
  Interventions: Other: Aerobic Exercise; Behavioral: Behavioral Treatment Program
- Control group (Active Comparator): A behavioral treatment program will be applied to the patients.
  Interventions: Behavioral: Behavioral Treatment Program

INTERVENTIONS:
Other: Aerobic Exercise — Aerobic Exercise training will be provided three days a week, 45 minutes a day, for 12 weeks. Patients will be subjected to submaximal aerobic exercise with rhythmic movements without equipment via video conference accompanied by a physiotherapist.
  Arms: Aerobic Exercise Group
Behavioral: Behavioral Treatment Program — Behavioral Treatment Program will be completed with an initial training period of 40 minutes, and subsequent control interviews of 20 minutes at four-week intervals.

SUMMARY:
The goal of this clinical trial is to investigate the effect of aerobic exercise (AE) on bladder functions and urinary system symptoms in women diagnosed with Diabetes Mellitus (DM) and suffered from Lower Urinary Tract Symptoms (LUTS). In the study, 44 individuals (35-55 age) were divided into two groups: Aerobic Exercise (AE) (n=22) and Control Group (n=22) by simple random method.

The main questions it aims to answer are:

* Is aerobic exercise effective on bladder functions in women diagnosed with Diabetes Mellitus and suffered from Lower Urinary Tract Symptoms?
* Is aerobic exercise effective on urinary tract symptoms in women diagnosed with Diabetes Mellitus and suffered from Lower Urinary Tract Symptoms?
* Is aerobic exercise effective on quality of life in women diagnosed with Diabetes Mellitus and suffered from Lower Urinary Tract Symptoms?

Intervention/treatment

* Control group individuals will be given a behavioral treatment program.
* Submaximal aerobic exercise training will be given to the AE group in addition to the behavioral treatment program.

DETAILED DESCRIPTION:
The goal of this clinical trial is to investigate the effect of aerobic exercise (AE) on bladder functions and urinary system symptoms in women diagnosed with Diabetes Mellitus (DM) and suffered from Lower Urinary Tract Symptoms (LUTS). In the study, 44 individuals (35-55 age) were divided into two groups: Aerobic Exercise (AE) (n=22) and Control Group (n=22) by simple random method. Bladder sensation (first sensation) and compliance from urodynamic evaluations will be taken as reference as the primary outcome measurement in treatment effectiveness.

* Control group individuals will be given a behavioral treatment program.
* Submaximal aerobic exercise training will be given to the AE group in addition to the behavioral treatment program.

AE training was provided three days a week, 45 minutes a day, for 12 weeks. The behavioral treatment protocol was completed with an initial training period of 40 minutes, and subsequent control interviews of 20 minutes at four-week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 35-55,
* Individuals who volunteer to participate in the study,
* Those diagnosed with Type II diabetes for 5 years or more and those diagnosed with LUTS

Exclusion Criteria:

* Stage 2 and more advanced pelvic organ prolapse,
* Urinary tract infection,
* Has had previous surgery for urinary incontinence and pelvic organ prolapse,
* Diagnosis of Cerebro Vascular Event (CVE) and dementia,
* Using A-blockers, antimuscarinics, antidepressants, diuretics and antihistamines,
* Individuals in menopause.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Bladder Compliance | 10 minutes (Change from Baseline at 12 weeks)
  Bladder compliance will be evaluated by urodynamics. With urodynamic evaluations, pathologies of the lower urinary system can be diagnosed and classified. Urodynamic examinations are performed in a suitable laboratory environment. First of all, a suitable sterile catheter is placed in the bladder and isotonic fluid is filled into it at a certain speed. In this way, the behavior of the bladder and its muscles during urine filling, pressure measurements and behavior during urination are examined. Bladder functions are evaluated with urodynamic evaluations. With the urodynamic evaluation will be performed by the clinician in the urology outpatient clinic compliance (ml/cmH2O) will be recorded.
Bladder Sensation | 10 minutes (Change from Baseline at 12 weeks)
  Bladder sensation will be evaluated by urodynamics. With urodynamic evaluations, pathologies of the lower urinary system can be diagnosed and classified. Urodynamic examinations are performed in a suitable laboratory environment. First of all, a suitable sterile catheter is placed in the bladder and isotonic fluid is filled into it at a certain speed. In this way, the behavior of the bladder and its muscles during urine filling, pressure measurements and behavior during urination are examined. Bladder functions are evaluated with urodynamic evaluations. With the urodynamic evaluation will be performed by the clinician in the urology outpatient clinic sensation (ml) will be recorded.

SECONDARY OUTCOMES:
Voiding Volume | 10 minutes (Change from Baseline at 12 weeks)
  Voiding volume will be evaluated by urodynamics. Urodynamic examinations are performed in a suitable laboratory environment. First of all, a suitable sterile catheter is placed in the bladder and isotonic fluid is filled into it at a certain speed. In this way, the behavior of the bladder and its muscles during urine filling, pressure measurements and behavior during urination are examined. Bladder functions are evaluated with urodynamic evaluations. With the urodynamic evaluation will be performed by the clinician in the urology outpatient clinic Voiding volume (ml) will be recorded.
Voiding Time | 10 minutes (Change from Baseline at 12 weeks)
  Voiding time will be evaluated by urodynamics. Urodynamic examinations are performed in a suitable laboratory environment. First of all, a suitable sterile catheter is placed in the bladder and isotonic fluid is filled into it at a certain speed. In this way, the behavior of the bladder and its muscles during urine filling, pressure measurements and behavior during urination are examined. Bladder functions are evaluated with urodynamic evaluations. With the urodynamic evaluation will be performed by the clinician in the urology outpatient clinic Voiding time (sec) will be recorded.
Maximum Bladder Capacity | 10 minutes (Change from Baseline at 12 weeks)
  Maximum bladder capacity will be evaluated by urodynamics. Urodynamic examinations are performed in a suitable laboratory environment. First of all, a suitable sterile catheter is placed in the bladder and isotonic fluid is filled into it at a certain speed. In this way, the behavior of the bladder and its muscles during urine filling, pressure measurements and behavior during urination are examined. Bladder functions are evaluated with urodynamic evaluations. With the urodynamic evaluation will be performed by the clinician in the urology outpatient clinic Maximum bladder capacity (ml) will be recorded.
Urine Maximum Flow Rate | 10 minutes (Change from Baseline at 12 weeks)
  Urine maximum flow rate will be evaluated by urodynamics. Urodynamic examinations are performed in a suitable laboratory environment. First of all, a suitable sterile catheter is placed in the bladder and isotonic fluid is filled into it at a certain speed. In this way, the behavior of the bladder and its muscles during urine filling, pressure measurements and behavior during urination are examined. Bladder functions are evaluated with urodynamic evaluations. With the urodynamic evaluation will be performed by the clinician in the urology outpatient clinic Maximum flow rate (ml/s) will be recorded.
Bladder Residual Volume | 10 minutes (Change from Baseline at 12 weeks)
  Bladder residual volume rate will be evaluated by urodynamics. Urodynamic examinations are performed in a suitable laboratory environment. First of all, a suitable sterile catheter is placed in the bladder and isotonic fluid is filled into it at a certain speed. In this way, the behavior of the bladder and its muscles during urine filling, pressure measurements and behavior during urination are examined. Bladder functions are evaluated with urodynamic evaluations. With the urodynamic evaluation will be performed by the clinician in the urology outpatient clinic Residual volume (cc) will be recorded.
Ultrasonography (USG) evaluation | 10 minutes (Change from Baseline at 12 weeks)
  Ultrasonography will be performed by the doctor using the measured thickest part of the bladder wall as reference. The wall thickness of the bladder (mm) will be noted when the bladder is empty and full. USG is a non-invasive imaging method that physicians routinely use to evaluate the urinary system.
Bladder Diary | Change from Baseline at 12 weeks
  48-hour bladder diary will be taken. The average of daily urination frequency numbers and daily fluid consumption amounts will be taken.
King's Health Questionnaire (KHQ) | Change from Baseline at 12 weeks
  It will be used to evaluate urinary system symptom severity and quality of life related to urinary system symptoms.The KHQ scale consists of two parts and 32 items. In the first part, there are two single-item questions about general health and quality of life. Again, in the first part, it consists of seven subheadings consisting of multiple items, including the individual's roles in daily life, physical condition, social situation, personal relationships, emotional problems, sleep/energy disorders, and violence measurements, and consists of 21 questions. The second part is a scale consisting of 11 questions that questions the presence of lower urinary tract symptoms and the severity of symptoms.Scoring on the Symptom Severity Scale ranges from 0 points (best) to 30 points (worst). In other KHQ subheadings, the scale scoring is 0 points (best) -100 points (worst). An increase in the score obtained from KHQ indicates a decrease in the quality of life.
Bristol Female Lower Urinary System Symptom Index (BFLUSSI) | Change from Baseline at 12 weeks
  It will be used to evaluate the Quality of Life Due to Lower Urinary System Symptoms.This scale includes storage functions (questions 1-4), excretory functions (questions 5-7), urinary incontinence (questions 8-12), sexual life (questions 13-14) and quality of life (questions 15-19). It consists of five sections with subheadings.
  The highest score that can be obtained from the survey is 71, while the lowest score is 0. A high score from the survey indicates that the severity of LUTS is high and sexual functions and quality of life are negatively affected.
HbA1c | Change from Baseline at 12 weeks
  HbA1c (blood glucose level) will be noted as a result of the blood evaluations taken by the clinician.
Patient Information Form | Change from Baseline at 12 weeks
  Patient information such as sociodemographic (age (year), occupation (employed/unemployed), education (literate/primary school/high school/university/graduate school), marital status (married/single), number of births (n), type of delivery (vaginal/caesarean section) and physical (height (m), weight (kg), BMI (kg/m2),constipation (, type 2 DM duration (year)) will be noted. Personal habits (liquid consumption habits (ml), number of urinations per day (n)) will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Bengisu TÜFEKÇİ, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No